CLINICAL TRIAL: NCT05281666
Title: Suture Repair of Lacerations in the Emergency Department: Comparison Between Absorbable and Non-absorbable Suture Material
Brief Title: Suture Repair of Lacerations in the ED: Comparison Between Two Suture Materials
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study closed due to recruitment problems
Sponsor: Kenneth Taylor, M.D. (Other)
Responsible Party: Sponsor-Investigator, Kenneth Taylor, M.D., Professor of Orthopaedics and Rehabilitation, Milton S. Hershey Medical Center
Organization: Milton S. Hershey Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00019465
Record Dates: First submitted 2022-03-07; First posted 2022-03-16 (Actual); Last update posted 2025-05-18 (Actual); Status verified 2025-05

CONDITIONS: Laceration of Hand; Laceration of Forearm
Keywords: laceration; wound; absorbable; non-absorbable; hand; forearm
MeSH Terms: conditions — Lacerations; Wounds and Injuries

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to either absorbable versus non-absorbable sutures and compared
Masking Description: No masking. Both participant and care providers will know group assignment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Absorbable Surgical Gut Suture (Active Comparator): Ethicon Chromic Surgical Gut Suture Is an absorbable, sterile surgical suture composed of purified connective tissue (mostly collagen) derived from either the serosal layer of beef (bovine) or the submucosal fibrous layer of sheep (ovine) Intestines. Surgical Gut Suture is Indicated for use In general soft tissue approximation and/or ligation, including use In ophthalmic procedures, but not for use in cardiovascular and neurologic tissues.
  Interventions: Device: Absorbable Surgical Gut Suture material
- Non-absorbable Nylon Suture (Active Comparator): Ethicon ETHILON* nylon suture is a nonabsorbab\e, sterile surgical monofi\ament suture composed of the long-chain aliphatic polymers Nylon 6 and Nylon 6,6. ETHILON sutures are dyed black or green to enhance visibility in tissue. The suture is also available undyed (clear). ETHILON suture is indicated for use in general soft tissue approximation and/or ligation, including use in cardiovascular, ophthalmic and neurological procedures.
  Interventions: Device: Non-absorbable Nylon Suture Material

INTERVENTIONS:
Device: Absorbable Surgical Gut Suture material — Participants with lacerations below the level of the forearm that meet inclusion criteria and are consented and randomized to this group will undergo washout and laceration repair using absorbable surgical gut suture material. They will be sent home with antibiotics. They will be asked to return to the outpatient hand clinic at 2, 6, and 12 weeks follow-up. Their wound will be assessed by a single observer, utilizing the POSAS and VAS.
  Arms: Absorbable Surgical Gut Suture
Device: Non-absorbable Nylon Suture Material — Participants with lacerations below the level of the forearm that meet inclusion criteria and are consented and randomized to this group will undergo washout and laceration repair using non-absorbable nylon gut suture material. They will be sent home with antibiotics. They will be asked to return to the outpatient hand clinic at 2, 6, and 12 weeks follow-up. Their sutures will be removed at the 2-week follow-up visit. Their wound will be assessed by a single observer, utilizing the POSAS and VAS.
  Arms: Non-absorbable Nylon Suture

SUMMARY:
This study aims to determine whether the use of non-absorbable (i.e. nylon) versus absorbable (i.e. chromic gut) sutures in traumatic hand lacerations affects wound healing, patient perception, and development of complications.

DETAILED DESCRIPTION:
There has been limited data published on suture type in traumatic hand wounds. The only study we found in our literature review was a retrospective study comparing vicryl vs. nylon suture and found no difference in scar appearance, tenderness, retraction, or complications as far as 6 months after repair (2). There have been no prospective studies on this topic. The theoretical advantage of absorbable suture for these wounds is they do not require suture removal, thereby removing the discomfort of suture removal as well potentially decreasing the burden of follow-up.

At the Penn State Health Hershey Medical Center, either suture choice included in this study is considered standard of care and is routinely used. Selection as to whether absorbable or non-absorbable suture is used is based on the preference and discretion of the resident and attending surgeon involved in the patient care. As such, if a patient were to present to the emergency department with a forearm or hand laceration and hand surgery were consulted, regardless of whether the patient opts to participate in this research study, their laceration would be repaired with either absorbable or non-absorbable suture depending on provider preference and the patient would be scheduled follow-up.

There have been multiple prospective clinical trials on suture type in the context of planned surgical incisions, specifically carpal tunnel release, with variable outcomes. One clinical trial looking at a total of 40 incisions found no difference in pain, tenderness, inflammation, or outcomes postoperatively (3). Certain clinical trials favored non-absorbable sutures, reporting a higher rate of infection (4) or inflammation (5) with vicryl suture as compared to non-braided, non-absorbable sutures. On the other hand, other clinical trials favored absorbable sutures, describing reduction in pain scores (6) and pain associated with absorbable suture removal in the setting of other equivalent outcomes (7).

The purpose of the study is to evaluate the use of absorbable and non-absorbable suture material in hand lacerations repaired in the Penn State Health Milton S. Hershey Emergency Department.

ELIGIBILITY:
Inclusion Criteria:

* Subject seen in PSHMC Emergency Department for hand or forearm lacerations (i.e. laceration below the level of the elbow) that require suture repair, in which Hand Surgery is consulted
* CDC surgical wound classification grades I-IV
* Age >18 years of age
* Gender: male or female (non-pregnant)
* Fluent in written and spoken English
* Subject is able to provide voluntary, written informed consent
* Subject, in the opinion of the clinical investigator, is able to understand the clinical investigation and is willing to perform all study procedures and follow-up visits
* Non-Prisoners

Exclusion Criteria:

* Known allergy to suture material
* History of immunosuppression (i.e. concurrent chemotherapy, steroid use or immunomodulatory therapy)
* History of diabetes mellitus
* Pregnancy
* Current Tobacco use
* Age < 18 years old
* Previous skin laceration at same location
* History of previous hypertrophic or keloid scar
* Concurrent tendon, nerve or bone injury requiring trip to the operating room
* Non-English speaking patients
* Cognitive impairment
* Prisoners

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2022-08-23 (Actual); Primary Completion 2025-05-06 (Actual); Study Completion 2025-05-06 (Actual)

PRIMARY OUTCOMES:
Change in wound healing using the Patient and Observer Scar Assessment Scale (POSAS) | 12 weeks
  Patients return to the practice site at 2 weeks, 6 weeks, and 12 weeks after their initial visit to the Emergency Department

SECONDARY OUTCOMES:
Patient reported pain using the Visual Analog Scale (VAS) | 12 weeks
  Patients return to the practice site at 2 weeks, 6 weeks, and 12 weeks after their initial visit to the Emergency Department

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth Taylor, MD, Principal Investigator — Penn State Health Milton S Hershey Medical Center
Locations (1):
- Penn State Health Milton S. Hershey Medical Center, Hershey, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Draaijers LJ, Tempelman FR, Botman YA, Tuinebreijer WE, Middelkoop E, Kreis RW, van Zuijlen PP. The patient and observer scar assessment scale: a reliable and feasible tool for scar evaluation. Plast Reconstr Surg. 2004 Jun;113(7):1960-5; discussion 1966-7. doi: 10.1097/01.prs.0000122207.28773.56. PMID 15253184
- [Background] Shetty PC, Dicksheet S, Scalea TM. Emergency department repair of hand lacerations using absorbable vicryl sutures. J Emerg Med. 1997 Sep-Oct;15(5):673-4. doi: 10.1016/s0736-4679(97)00147-9. PMID 9348057
- [Background] Kharwadkar N, Naique S, Molitor PJ. Prospective randomized trial comparing absorbable and non-absorbable sutures in open carpal tunnel release. J Hand Surg Br. 2005 Feb;30(1):92-5. doi: 10.1016/j.jhsb.2004.10.009. PMID 15620502
- [Background] Menovsky T, Bartels RH, van Lindert EL, Grotenhuis JA. Skin closure in carpal tunnel surgery: a prospective comparative study between nylon, polyglactin 910 and stainless steel sutures. Hand Surg. 2004 Jul;9(1):35-8. doi: 10.1142/s0218810404002017. PMID 15368623
- [Background] Erel E, Pleasance PI, Ahmed O, Hart NB. Absorbable versus non-absorbable suture in carpal tunnel decompression. J Hand Surg Br. 2001 Apr;26(2):157-8. doi: 10.1054/jhsb.2000.0545. PMID 11281671
- [Background] Hansen TB, Kirkeby L, Fisker H, Larsen K. Randomised controlled study of two different techniques of skin suture in endoscopic release of carpal tunnel. Scand J Plast Reconstr Surg Hand Surg. 2009;43(6):335-8. doi: 10.1080/02844310902955763. PMID 19995253
- [Background] Freshwater MF. Theopold C, Potter S, Dempsey M, O'Shaughnessy M. A randomised controlled trial of absorbable versus non-absorbable sutures for skin closure after open carpal tunnel release. J Hand Surg Eur. 2012; 37: 350-3. J Hand Surg Eur Vol. 2012 Sep;37(7):705; author reply 705-6. doi: 10.1177/1753193412454501. No abstract available. PMID 22879647
- [Background] Onyekwelu I, Yakkanti R, Protzer L, Pinkston CM, Tucker C, Seligson D. Surgical Wound Classification and Surgical Site Infections in the Orthopaedic Patient. J Am Acad Orthop Surg Glob Res Rev. 2017 Jun 13;1(3):e022. doi: 10.5435/JAAOSGlobal-D-17-00022. eCollection 2017 Jun. PMID 30211353